CLINICAL TRIAL: NCT04382521
Title: A Text Message Intervention to Promote Health Behaviors in Cardiac Risk Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Director of Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019P003495
Record Dates: First submitted 2020-04-25; First posted 2020-05-11 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hyperlipemia; Hypertension; Type2 Diabetes
Keywords: text message intervention; health behavior change; positive psychology
MeSH Terms: conditions — Hyperlipidemias; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message Intervention (TMI) (Experimental): Participants in the TMI condition will receive daily text messages through an adaptive algorithm plus separate twice-weekly tailored messages focused on a specific health goal.
  Interventions: Behavioral: Text Message Intervention
- Wait-list Control Group (WLC) (Other): Waitlist Control group participants will begin to receive the full 12-week Text Message Intervention (with all components, e.g., phone check-ins) after completing follow-up assessments at Weeks 12 and 24. Participants in this group will receive no text messages or other study-specific interventions during the first 24 weeks of the study.
  Interventions: Behavioral: Text Message Intervention

INTERVENTIONS:
Behavioral: Text Message Intervention — Participants will undergo a three component intervention consisting of (1) daily, adaptive text messages related to Positive Psychology or health behaviors, (2) twice weekly text messages related to a specific health behavior goal, and (3) three brief check-ins (at baseline, week 4, and week 8 of the intervention) with a study staff member to discuss progress towards health behavior goals. During the brief check-ins, the study staff member will inquire about: (1) medical conditions, (2) adherence gaps, (3) personal health goals (including weight goals), (4) motivation, self-efficacy, and barriers to reaching health goals, (5) preferred activity types (e.g., walking), and (6) sources of sedentary time (e.g., computer, TV). This information will be added to the algorithm for each individual and we will deliver tailored daily text messages for our participants.

SUMMARY:
This is a randomized pilot trial to examine the feasibility, acceptability, and preliminary efficacy of an adaptive text message intervention (TMI) to promote well-being and health behavior adherence in 60 patients with two or more cardiac risk conditions (hypertension, type 2 diabetes, or hyperlipidemia).

DETAILED DESCRIPTION:
The investigators have developed an adaptive text message intervention (TMI) that uses participant feedback for individual messages and progress towards health goals to deliver increasingly personalized positive psychology (PP) and health behavior text messages over time. The investigators aim to examine its feasibility, acceptability, and preliminary efficacy in a randomized, controlled pilot trial in 60 adults with two or more cardiac risk conditions (hypertension, type 2 diabetes, or hyperlipidemia).

ELIGIBILITY:
Inclusion Criteria:

* Cardiac risk conditions. Participants will have two or more of hypertension, type-2 diabetes, and hyperlipidemia. Patients will have met 2+ of 2017 AHA-ACC criteria for hypertension (SBP ≥130, DBP ≥80), 2018 ADA criteria for type-2 diabetes (e.g., A1C ≥6.5%), and 2013 AHA-ACC criteria for hyperlipidemia (e.g., LDL cholesterol ≥190), via medical record review, with confirmation by healthcare providers as needed.
* Low physical activity or elevated sedentary leisure time (SLT). Low activity will be defined as ≤150 minutes/week of moderate to vigorous activity (MVPA), which is an ADA-recommended level of MVPA; elevated SLT will be ≥120 min/day, which is linked to adverse medical health. As initial screens for both MVPA and SLT, we will use the International Physical Activity Questionnaire (IPAQ). Patients reporting ≤150 min/week of MVPA or ≥120 min/day of SLT will wear accelerometers for 10 days to confirm low MVPA/high SLT (patients will indicate their leisure time hours to allow assessment of SLT during those hours).
* Suboptimal diet. Participants must also report either fewer than 5 daily servings of fruit/vegetables (measured by the Behavioral Risk Factor Surveillance System's [BRFSS] Fruit and Vegetable Consumption Module) or have a score of ≥70 on the MEDFICTS scale for fat/cholesterol intake, representing high risk. We will require diet and activity deficits to ensure that a broad range of messages will be relevant to every participant as we explore the utility of individual messages and patterns of message selection in this initial study.
* Ability to receive text messages. Participants must have a cellular phone that receives texts and that they use at least daily. We will remunerate them the cost of receiving the messages as needed.
* Ability to read in English or Spanish. Text messages will be available in English and Spanish.

Exclusion Criteria:

* Existing coronary artery disease (CAD; diagnosed via cardiac catheterization using standard coronary artery stenosis definitions or prior ACS).
* An unrelated condition limiting physical activity.
* Participation in programs focused on cardiac prevention or well-being (e.g., cardiac rehabilitation).
* A cognitive disturbance precluding participation or informed consent, assessed using a six-item screen designed to assess suitability for research participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion of messages correctly delivered | 12 weeks
  Proportion of adaptive TMI messages correctly selected/sent will be included as a measure of feasibility.
Rates of feedback to individual text messages | 12 weeks
  Rates of feedback to individual text messages will be included as a measure of feasibility.
Participant's mean ratings of message utility to measure acceptability of the text-message intervention | 12 weeks
  0-10 Likert scale score regarding the utility of that day's text message

SECONDARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) Score | Baseline, 12 weeks and 24 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect. (Range: 10-50). Higher scores indicate higher levels of positive affect. The measure will be used at baseline, 12 weeks and 24 weeks.
Change in Life Orientation Test-Revised Score | Baseline, 12 weeks and 24 weeks
  Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism. (Range: 0-24) Higher scores indicate higher levels of optimism. The measure will be used at baseline, 12 weeks and 24 weeks.
Change in General Self-Efficacy Scale score | Baseline, 12 weeks and 24 weeks
  The General Self-Efficacy Scale is a self-report measure of self-efficacy. The total score ranges from 10-40, with a higher score indicating more self-efficacy.
Change in HADS-A Score | Baseline, 12 weeks and 24 weeks
  The anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A) will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound anxiety assessment in medically-ill patients. (Range: 0-21) Higher scores indicate higher levels of anxiety. The measure will be used at baseline, 12 weeks, and 24 weeks.
Change in HADS-D Score | Baseline, 12 weeks and 24 weeks
  The depression subscale of the Hospital Anxiety and Depression Scale (HADS-D) will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood assessment in medically-ill patients.(Range: 0-21). Higher scores indicate worse outcome (i.e. greater levels of depression). The measure will be used at baseline, 12 weeks, and 24 weeks.
Change in Multidimensional Health Locus of Control Score | Baseline, 12 weeks and 24 weeks
  This is an 18-item instrument that measures three dimensions of locus of control. It assesses people's beliefs that their health is or is not determined by their own behavior. The survey has three subscales: internality of health locus of control, powerful other locus of control, and chance locus of control. All items are measured on a 6-point Likert scale, and our main subscale of interest will be internal locus of control, which will be a sum of scores from questions 1,6,8,12,13,17 (range: 6-36). Higher scores indicate higher locus of control.
Change in Multidimensional Scale of Perceived Social Support Score | Baseline, 12 weeks and 24 weeks
  The MSPSS is a 12-item scale designed to measure perceived social support from three sources: Family, Friends, and a Significant Other. It is rated on a 7-point likert scale, ranging from 1 "very strongly disagree" to 7 "very strongly agree." Each subscale score can range from 4 to 28. Items are summed, and a total score is also calculated and ranges from 12 to 84. Higher subscale and total scores indicate high levels of perceived social support.
Change in MEDFICTS score | Baseline, 12 weeks and 24 weeks
  MEDFICTS is a screening instrument for dietary fat to assess adherence to the Adult Treatment Panel (ATP) III Therapeutic Lifestyle Changes (TLC) diet. The test measures the intake of meats, eggs, dairy, fried foods, fats in baked goods, convenience foods, table fats, and snacks. Higher scores indicate higher fat consumption.
Change in Behavioral Risk Factor Surveillance System [BRFSS] Fruit and Vegetable Consumption Module | Baseline, 12 weeks and 24 weeks
  The CDC's BRFSS Fruit and Vegetable Module is a brief questionnaire about frequency of eating different types of fruits and vegetables. It assesses the frequency of consumption of 100% fruit juice, fruit, beans (legumes), dark green vegetables, orange vegetables, and other vegetables over the past month. The outcome measure is the number of fruits or vegetables consumed per day.
Change in Moderate to vigorous physical activity (minutes) measured via accelerometer | Baseline, 12 weeks and 24 weeks
  Measured by Actigraph accelerometer, in minutes per day.
Change in physical activity (steps) measured via accelerometer | Baseline, 12 weeks and 24 weeks
  Measured by Actigraph accelerometer, in number of steps per day.
Change in sedentary time measured via accelerometer | Baseline, 12 weeks and 24 weeks
  Measured by Actigraph accelerometer, in minutes per day.
Change in self-report physical activity time measured by International Physical Activity Questionnaire | Baseline, 12 weeks and 24 weeks
  Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assess the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. The measure will be used at baseline, 12 weeks, and 24 weeks.
Change in physical function measured by PROMIS 20-item | Baseline, 12 weeks and 24 weeks
  Measured by the 20-item short form of the Patient-Reported Outcomes Measurement Information System (PROMIS), a well-validated measure of physical function that is highly responsive to changes in a patient's physical function status (Range: 20-100). Higher scores indicate better physical function.
Change in physical function measured by 6-minute test | Baseline, 12 weeks and 24 weeks
  The 6-minute walk test is a test to measure participant's functional capacity, assessing distance walked in meters in 6 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celano CM, Healy BC, Jacobson LH, Bell M, Carrillo A, Massey CN, Chung WJ, Legler SR, Huffman JC. An adaptive text message intervention to promote psychological well-being and reduce cardiac risk: The Text4Health controlled clinical pilot trial. J Psychosom Res. 2024 Feb;177:111583. doi: 10.1016/j.jpsychores.2023.111583. Epub 2023 Dec 30. PMID 38171212